CLINICAL TRIAL: NCT01806636
Title: Post Market Observational, Prospective, Multi-center Registry Using the PneumRx, Inc. Lung Volume Reduction Coil (LVRC) System
Brief Title: Post Market Observational, Prospective, Multi-center Study
Status: Terminated | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: PneumRx, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN0014
Record Dates: First submitted 2013-02-17; First posted 2013-03-07 (Estimated); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Emphysema
Keywords: Coil; RePneu; PneumRx; LVRC
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment: Patients treated with PneumRx Coil System
  Interventions: Device: PneumRx Coil System

INTERVENTIONS:
Device: PneumRx Coil System
  Other Names: RePneu; LVRC

SUMMARY:
This registry is a post market observational, prospective, multi-center registry.

It is designed to evaluate patient experience with the endobronchial coil system for the relief of the emphysema symptoms and the continued collection of safety and effectiveness data on this CE Mark product.

ELIGIBILITY:
Inclusion and exclusion criteria in the Registry are based on CE Mark approved indication and approved Instructions for Use. Patients enrolled and treated in the Registry study should meet the requirements of the PneumRx Endobronchial Coil System Instructions for Use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients diagnosed with homogeneous or heterogeneous emphysema who are appropriate for Coil treatment based on the CE-Mark Approved IFU and who have been scheduled for treatment with the RePneu procedure will be eligible to participate in the Registry. If they agree and sign a consent form, they will then become study participants.
Sampling Method: Probability Sample
Enrollment: 1275 (Actual)
Dates: Start 2013-05; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Changes in Quality of Life (QOL) measures | 6 months and yearly up to three years post treatment 1

SECONDARY OUTCOMES:
Changes in Pulmonary Function and Exercise Capacity test results | 6 months and yearly up to three years post treatment 1
Safety including any device malfunction or failure(s) | 6 months and yearly up to three years post treatment 1

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hetzel, Prof., Principal Investigator — Krankenhaus vom Roten Kreuz; Christian Schumann, MD, Principal Investigator — Klinikenverbund Kempten-Oberallgäu
Locations (73):
- Otto-Wagner-Spital, Vienna, Austria
- Rigshospitalet Copenhaven, Copenhagen, Denmark
- Germany (51):
  - Hochtaunus-Kliniken, Klinik für Pneumolog und Onkologie, Bad Homburg
  - Charité Campus Mitte, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - Gemeinschaftskrankenhaus Havelhöhe, Berlin
  - Helios Klinikum Emil von Behring, Berlin, Berlin-Zehlendorf
  - Universitätsklinikum Bonn, Bonn
  - Ev. Krankenhaus Göttingen-Weende, Bovenden
  - DRK Klinik am Bürgerpark, Bremerhaven
  - Kreiskliniken Altötting-Burghausen, Burghausen
  - St. Marien-Hospital, Cologne
  - Schwarzwald-Baar-Klinikum, Donaueschingen
  - Klinik Donaustauf, Donaustauf
  - Medizinische Klinik Nord, Dortmund
  - HELIOS Klinikum Duisburg, Duisburg
  - Johanniter KH Duisburg Rheinhausen, Duisburg
  - Pneumologische Klinik Waldhof Elgershausen, Elgershausen
  - Ruhrlandklinik, Essen
  - Bethanien Krankenhaus, Frankfurt am Main
  - St. Elisabethen Krankenhaus, Frankfurt am Main
  - Klinikum Fürth, Fürth
  - Asklepios-Klinikum Gauting, Gauting
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Universitätsmedizin Greifswald, Greifswald
  - Universitätsklinikum Halle, Halle
  - Diakoniekrankenhaus Halle, Halle
  - Uniklinik Eppendorf, Hamburg
  - Asklepios Klinik Barmbeck, Hamburg
  - Asklepios, Harburg
  - Lungenklinik, Hemer
  - Lungenfachklinik Immenhausen, Immenhausen
  - Klinikverbund Kempten-Oberallgäu, Kempten
  - Marienhof Koblenz, Koblenz
  - HELIOS Klinikum Krefeld, Krefeld
  - Lungenklinik Lostau, Lostau
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitätsklinikum Magdeburg, Magdeburg
  - Katholisches Klinikum Mainz, Mainz
  - Krankenhaus Martha-Maria, München
  - Städt. Klinikum München-Harlaching, München
  - Städt. Klinikum München-Bogenhausen, München
  - Ruppiner Kliniken GmbH, Neuruppin
  - Brüderkrankenhaus St. Josef Paderborn, Paderborn
  - Universitätsklinikum, Regensburg
  - RoMed Klinikum Rosenheim, Rosenheim
  - Helios Kliniken Schwerin, Schwerin
  - Krankenhaus Bethanien Solingen, Solingen
  - Krankenhaus vom Roten Kreuz, Stuttgart
  - Universitätsklinikum Ulm, Ulm
  - Saarland Heilstätten GmbH, Völklingen
  - Petrus-Krankenhaus, Wuppertal
  - Medizinisches Zentrum Städte Region Aachen GmbH, Würselen
- Spain (6):
  - Centro Médico Teknon, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Universitario Quirón, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Quiron, Málaga
  - Hospital Universitario y Politécnico La Fe, Valencia
- Switzerland (7):
  - Inselspital, Bern
  - Hôpitaux Universitaires de Genève (HUG), Geneva
  - CHUV, Lausanne
  - L'hôpital Neuchâtelois - Pourtalès, Neuchâtel
  - Kantonsspital Sankt Gallen, Sankt Gallen
  - Lungenzentrum Hirslanden, Zurich
  - UniversitätsSpital Zürich, Zurich
- United Kingdom (7):
  - Heartlands Birmingham, Birmingham
  - Bristol Royal Infirmary, Bristol
  - Leicester Royal Infirmary, Leicester
  - Guy's and St Thomas' Hospital, London
  - Royal Brompton Hospital, London
  - Royal Preston Hospital, Preston
  - Southampton General Hospital, Southampton